CLINICAL TRIAL: NCT07056296
Title: Efficiency of a New Versatile Three-Way Maxillary Expander Versus Modified Fan Expander for Maxillary Arch Expansion in Cleft Lip and Palate Patients: A Randomized Controlled Trial
Brief Title: Efficiency of Two Maxillary Expanders for Maxillary Arch Expansion in Bilateral Cleft Lip and Palate Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-Rec ID 052316
Record Dates: First submitted 2025-06-15; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2023-05

CONDITIONS: Bilateral Cleft Lip and Palate; Maxillary Expansion
Keywords: Bilateral cleft lip and palate; Expansion; Premaxilla; Three-dimensional expansion; Fan expander; Three- way expander

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three-way iMini Hyrax group (Experimental): For group (A) cases, a custom-made Three-way palatal expansion appliance will be made. The appliance design will be composed of: Orthodontic bands on first permanent molars. Three mini-expansion screws with two break resistant retention legs, oriented as follows: a transverse screw and bilateral sagittal screws.
  Interventions: Device: 3D Maxillary Expansion with 3 expansion screws
- Fan Expander group (Active Comparator): For group (B) cases, a custom-made modified Fan palatal expansion appliance will be made. The appliance design will be composed of: Orthodontic bands on first permanent molars. A fan expansion screw with break resistant retention legs with soldered finger springs just palatal to the premaxilla.
  Interventions: Device: 3D Maxillary Expansion using modified Fan expander with springs

INTERVENTIONS:
Device: 3D Maxillary Expansion with 3 expansion screws — In patients requiring maxillary expansion, after randomization and allocation for each to receive which expander, appliance will be cemented. In the 3-way group (A), 3 screw activations will be delivered by the care giver to expand the maxillary arch in 3D manner correcting the collapsed arch anteriorly.
  Other Names: 3-way expander; Group (A)
  Arms: Three-way iMini Hyrax group
Device: 3D Maxillary Expansion using modified Fan expander with springs — For the fan expander with palatal springs (B) , spring activation will be done by the operator after cemenation intraorally, then the care giver too will just activate one fan screw. Also 3D expansion evaluation was done.
  Other Names: Fan expander; Group (B)
  Arms: Fan Expander group

SUMMARY:
This randomized controlled trial is designed to compare between Fan expander with palatal springs appliance vs three-way expander regarding the their effectiveness in maxillary expansion in patients with bilateral cleft

DETAILED DESCRIPTION:
The study provides three-dimensional expansion for cleft lip and palate patients. Patients with repaired cleft lip and/or palate have maxillary deficiency and hypoplasia in the three planes of space. Most cases have a normal buccolingual occlusal relation in the molar region between upper and lower jaws, while they manifest arch constriction at the anterior inter-canine width area as well as premaxillary collapse and anterior crossbite. Conventional expansion appliances address only the transverse discrepancy requiring a further step to re-align the premaxilla. So, the aim of the study is to compare the efficiency and the effects of the new design of the three-way palatal expander and the modified fan expander in maxillary arch development in cleft lip and palate patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age ranging from 8 to 15 years old.
* Patients with bilateral cleft lip and palate.
* Patients with repaired cleft lip and / or palate.
* Patients with fully erupted upper permanent 1st molars.
* Patients in the late mixed or early permanent dentition with tapered maxillary arch, requiring palatal expansion as part of their treatment.
* Patient's stage of cervical vertebral maturation before or at the growth spurt (CS1-CS4).

Exclusion Criteria:

* Patients with syndromic cleft lip and palate.
* Patients with very bad oral hygiene and active periodontal disease.
* Vulnerable groups

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Maxillary arch development in Anteroposterior dimension | [Time Frame: 6 - 12 months]
  Anterior expansion of the premaxilla in the sagittal plane measured through lateral Cephalograms

SECONDARY OUTCOMES:
Inter-canine width expansion in the transverse plane | [Time Frame: 6- 12 months]
  Inter-canine width expansion in the transverse plane measured on Digital dental models.
Dental changes with expansion | [Time Frame: 6- 12 months]
  Amount of dental tipping occurring with expansion and amount of expansion and distal movement of maxillary molars

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, Ain Shams University, Cairo, Abbaseya, Egypt

IPD SHARING:
Plan to Share IPD: No